CLINICAL TRIAL: NCT07348406
Title: Effects of Pecans on Brain Health in Older Americans With Mild Cognitive Impairment: Gut-brain Axis
Brief Title: Snacks and Brain Health
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-FY2026-58
Record Dates: First submitted 2025-12-29; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Cognitive Assessment; Psychological Function; GI Health
Keywords: neuroinflammation; gut microbiome; fMRI
MeSH Terms: conditions — Neuroinflammatory Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pecan (Active Comparator): 2.0 oz pecans daily for 3 months
  Interventions: Biological: Pecan snack
- Pretzel (Placebo Comparator): 3.5 oz pretzel snack daily for 3 months
  Interventions: Biological: Pretzel snack

INTERVENTIONS:
Biological: Pecan snack — Pecan
  Arms: Pecan
Biological: Pretzel snack — Pretzel snack
  Arms: Pretzel

SUMMARY:
This project will investigate whether daily snack consumption can improve memory, mood, and overall brain function in people with cognitive impairment. Sixty participants, aged 50 and older, with cognitive impairment, will be randomly assigned to eat snacks, either pecans or pretzels, for three months. Researchers will also study how snacks (pecans and pretzels) may influence the body, including changes in gut bacteria, blood markers of inflammation, and signals that connect the gut and the brain.

ELIGIBILITY:
Inclusion Criteria:

* men and women > 50 years-old
* self-reported IQCODE (informant questionnaire on cognitive decline in the elderly) average score < 4.5
* self-reported significant functional impairment (related to cognitive impairment) in basic or advanced activities of daily living as evidenced by the Activities of Daily Living (ADLs) questionnaire. If answers to at least one endorsement in the "NO, dependence due to memory concerns".
* Stable medications (≥ 12-week unchanged dose before baseline) with no planned changes during trial.
* habitually consume less than two servings (2 ozs = 1/4 cup) of nuts or nut spreads per week
* willing to accept randomization

Exclusion Criteria:

* reported nut allergy or intolerance
* self-reported untreated hypothyroidism, severe liver disease, or end-stage chronic kidney disease
* heavy alcohol drinker: in the past 3 months: men ≥14 drinks/week or women ≥7 drinks/week
* recent (<1 month) appearance of diarrhea or hematochezia before study intervention begins. Rationale: A one-month waiting period after diarrhea or hematochezia (blood in stool) is recommended for a gut microbiome test to ensure the results accurately reflect the state and microbial composition, since diarrhea and hematochezia can significantly alter the gut environment and skew test results.
* recent (<1 month) exposure to antibiotics before study intervention begins. Rationale: A one-month waiting period after antibiotics is recommended for a gut microbiome test because it allows the microbial community time to recover and reach a more stable state, ensuring a more accurate and representative snapshot of the gut microbiome composition, since antibiotic usage can significantly reduce microbial diversity.
* Self-reported unstable GI disorder
* likeliness of moving during the trial, lack of transportation, or unavailability at sample collection times

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
fMRI measures | baseline and after 3 months
  connectivity of amygdala seed regions and broader bilateral mPFC using fMRI

SECONDARY OUTCOMES:
NACC Uniform Data Set | baseline and after 3 months
  overall neurocognitive functioning
Wisconsin Card Sorting Test | baseline and after 3 months
  Cognition
California Verbal Learning Test | baseline and after 3 months
  Memory and verbal learning
Clock Draw Test | baseline and after 3 months
  Visuospatial functioning
TRAILS A and B | baseline and after 3 months
  neuropsychological function
Geriatric Depression Scale (GDS-15) | baseline and after 3 months
  Depression assessment
Beck Anxiety Inventory (BAI) | baseline and after 3 months
  Anxiety assessment
fecal zonulin concentration by ELISA | baseline and after 3 months
  Intestinal permeability marker
gut microbiome | baseline and after 3 months
  fecal microbiome composition using 16S RNA sequencing
fecal metabolites | baseline and after 3 months
  untargeted fecal metabolites by LC-MS analysis
neuroinflammation gene | baseline and after 3 months
  whole blood neuroinflammation gene profiles

CONTACTS AND LOCATIONS:
Overall Officials: Chwan-Li (Leslie) Shen, PhD, Principal Investigator — Texas Tech University Health Sciences Center School of Medicine
Locations (1):
- Texas Tech University Health Sciences Center, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available due to HIPAA regulation.